CLINICAL TRIAL: NCT04027972
Title: Pharmacokinetics of Neostigmine and Glycopyrrolate After Intravenous and Transcutaneous Administration by Iontophoresis
Brief Title: Pharmacokinetics of Neostigmine and Glycopyrrolate
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chris Cardozo, Principal Investigator, James J. Peters Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOR-18-16
Record Dates: First submitted 2019-07-19; First posted 2019-07-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries; Constipation; Fecal Incontinence; Neurogenic Bowel
Keywords: Neostigmine; Glycopyrrolate; Transdermal; Intravenous; Pharmacokinetic; Constipation; Bowel Control; Mass Spectroscopy; Stool Incontinence
MeSH Terms: conditions — Spinal Cord Injuries; Constipation; Fecal Incontinence; Neurogenic Bowel; Encopresis | interventions — Glycopyrrolate; Iontophoresis

STUDY DESIGN:
Intervention Model Description: Same group receives all 2 treatments but in a randomized order after the IV phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Primary (Experimental): 6 Subjects will receive all 4 types of medication administration in random sequence
  Interventions: Drug: Combination of Neostigmine and Glycopyrrolate; Device: I-Box by Dynatronics

INTERVENTIONS:
Drug: Combination of Neostigmine and Glycopyrrolate — Intravenous or transdermal
Device: I-Box by Dynatronics — Electric field conducting drugs through the skin without compromising its integrity
  Other Names: Iontophoresis

SUMMARY:
A group of 6 able-bodied healthy volunteers will receive Neostigmine (NEO) and Glycopyrrolate (GLY) intravenously and via 2 methods of Iontophoresis (ION): one-patch and two-patch administration, with subsequent blood draws over 1 hour in order to measure the pharmacokinetic behavior of the drugs in-vivo.

DETAILED DESCRIPTION:
The maximum dose of NEO is limited to 10.0 mg and the dose of GLY to 2.0 mg per subject per administration. Subjects will be asked to arrive at the Spinal Cord Research Center at the JJP VAMC (Room 7A-13) on the day of their appointment. On Day 1, following the obtainment the subject's consent, filling out a MoCA cognitive assessment and establishing an IV access point, administration of the medications via IV will be performed. The study design will consist of a Day 1 visit to determine the pharmacokinetic profiles of the IV doses of NEO and GLY. During the second visit, at least 24 hours later, NEO (0.07 mg/kg) and GLY (0.014 mg/kg), applied separately to two patches, will be simultaneously delivered by transdermal administration by ION for 20 minutes. During the third and final visit, at least 24 hours following the second visit, a single patch containing 0.07 mg/kg of NEO and 0.014 mg/kg of GLY will be applied to the skin and delivered by transdermal administration by ION for 20 minutes..

Heart rate, bowel sounds, blood pressure and symptoms will be recorded at 0, 2, 4, 7, 10, 20, 40, 60 minutes of the initiation of the IV push and at 0, 10, 20, 40 and 60 minutes after the initiation of ION. Bowel evacuation time and time after the completion of delivery (by either ION or IV) will be recorded throughout the study visit, as described in Table 2. The subject will assume his/her normal bowel evacuation (BE) position until a bowel movement occurs; privacy draping and privacy will be provided at the time of BE. The subjects will be monitored for a minimum of 60 minutes. A minimum of two research personnel will be present during the study visit to record all of data and perform the tasks required.

After the start a 30 second IV push of NEO which will be followed by a NS flush (12 mL), and then a 30 second IV push of GLY which will be followed by a NS flush (12 mL), venous blood (2 mL) will be drawn into a gold-topped vial at 2, 4, 7, 10, 20, 40 and 60 minutes. Identical technique blood draws will be performed at 10, 20, 30, 40 and 60 minutes after the start of ION. Upon drawing, the blood will be placed in an ice bath and spun using a cooled centrifuge within 5 minutes of collection. Upon completion of 5 minutes of centrifugation, the resulting serum will be aliquoted into two separate vials, with equal volumes and labelled with date, time of draw, associated procedure, NEO or GLY testing destination and the subject's unique identifier. The transfer vials will be inserted into dry ice for at least 10 minutes, after which they will be placed into the -80 degrees Celsius freezer. Plasma levels of NEO and of GLY will be batched and measured at a later date. A file designating the tubes with random numbers associated with the draw times will be created for each subject to conceal the sequence of draw and to attempt the removal of possible bias during the measurement and recording of the concentrations of NEO and GLY (SUNY Downstate Albany Research Laboratory using GE LC-MRM detector).

Proposed Doses:

Day 1: 0.02 mg/kg NEO and 0.004 mg/kg GLY via IV

Day 2: 0.07 mg/kg NEO and 0.014 mg/kg GLY via ION (Two patch administration)

Day 3: 0.07 mg/kg NEO and 0.014 mg/kg GLY via ION (One patch administration)

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age 18-70 years

Exclusion Criteria:

* Previous adverse reaction or hypersensitivity to electrical stimulation,
* Known sensitivity to neostigmine or glycopyrrolate,
* History of mechanical obstruction of the GI or urinary tract,
* Myocardial infarction within 6 months of trial,
* Malignant and/or Uncontrollable Hypertension Defined by a blood pressure reading of 160/100 mmHg or higher with or without taking 3 or more different classes of anti-hypertensive medications,
* Organ damage (heart & kidney) and/or TIA-CVA as a result of hypertension,
* Known past history of coronary artery disease or bradyarrhythmia,
* Symptomatic orthostatic hypotension
* Deep brain stimulation
* Pregnancy (women who are sexually active and of childbearing potential must utilize a method of contraception and agree to maintain a contraceptive method until completion of the study),
* Lactating, nursing females
* Inability to provide informed consent signaled by MoCA cognitive test score of 20 or less,
* History of ingrown hair folliculitis,
* Concurrent illness and fever,
* Concurrent participation in a research study,
* VA employee.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of Neostigmine and Glycopyrrolate within 1 hour post-administration | Within Two Hours
  Measurement of serum concentration of Neostigmine and of Glycopyrrolate to determine pharmacokinetic profiles

SECONDARY OUTCOMES:
Presence or absence of headache, dry mouth, muscle twitching and abdominal cramps. | Within 1 hour of administration
  Determining safety of drug via presence or absence of headache, dry mouth, muscle twitching, and abdominal cramps as reported by the subjects

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Cardozo, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J Peters VA Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korsten MA, Lyons BL, Radulovic M, Cummings TM, Sikka G, Singh K, Hobson JC, Sabiev A, Spungen AM, Bauman WA. Delivery of neostigmine and glycopyrrolate by iontophoresis: a nonrandomized study in individuals with spinal cord injury. Spinal Cord. 2018 Mar;56(3):212-217. doi: 10.1038/s41393-017-0018-2. Epub 2017 Nov 8. PMID 29116244
- [Background] Korsten MA, Rosman AS, Ng A, Cavusoglu E, Spungen AM, Radulovic M, Wecht J, Bauman WA. Infusion of neostigmine-glycopyrrolate for bowel evacuation in persons with spinal cord injury. Am J Gastroenterol. 2005 Jul;100(7):1560-5. doi: 10.1111/j.1572-0241.2005.41587.x. PMID 15984982
- [Background] Chang JY, Locke GR 3rd, McNally MA, Halder SL, Schleck CD, Zinsmeister AR, Talley NJ. Impact of functional gastrointestinal disorders on survival in the community. Am J Gastroenterol. 2010 Apr;105(4):822-32. doi: 10.1038/ajg.2010.40. Epub 2010 Feb 16. PMID 20160713
- [Background] Sabiev A, Korsten MA, Bauman WA (2021) A Comparison among Three Skin Preparations for the Transdermal Delivery of Vitamin B12 by Iontophoresis: A Novel Approach to Determine Systemic Absorption. J Pharm Drug Deliv Res 10:3.

DOCUMENTS (1):
  • Informed Consent Form (2023-02-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT04027972/ICF_000.pdf